CLINICAL TRIAL: NCT06040645
Title: Outcomes of Urinary Incontinence Treatment in Primary Care: APP Co-Management and Electronic Consult
Acronym: OUTPACE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of California, Los Angeles (Other); University of Kansas (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jennifer Anger, Professor of Urology, Vice Chair of Research, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 806024
Record Dates: First submitted 2023-06-22; First posted 2023-09-15 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Urinary Incontinence
Keywords: Practice-based intervention; Patient-centered outcomes research; Disparities; Referrals; Quality of care indicators; Primary care
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electronic Consult (E-consult) (Experimental): In Arm 1, the investigators will implement an electronic referral system (electronic co-management), in which specialists will electronically review referrals and make additional recommendations if appropriate primary UI care was not provided.
  Interventions: Other: E-consult
- Advanced Practice Provider (APP) Co-management (Experimental): In Arm 2, Advanced Practice Provider (APP) co-management will reduce the burden of care on the PCPs by providing UI care, patient education, and assisting with patient self-management through dedicated televisits (APP co-management).
  Interventions: Other: APP Co-management

INTERVENTIONS:
Other: APP Co-management — To reduce additional burden of care on the PCPs, the investigators will incorporate Advanced Practices Providers into the patient education and self-management portion of care. The APPs will be trained together with the intervention physicians, but they will also undergo additional standardized training on patient education, UI knowledge, providing instruction on Kegel exercises, shared decision making, and self management.
  Patients will then be scheduled for a UI education and self-management session with the APP by telemedicine (video visit or telephone visit) within one month of their initial visit. For patients in need of an annual pelvic examination, and if the patient's PCP prefers to have the APP conduct the pelvic exam, a separate visit will be scheduled with the APP. A followup televisit will then be scheduled within three months of the initial APP visit, in order to assess the outcome of non-surgical treatment and determine if a specialist referral is indicated.
  Arms: Advanced Practice Provider (APP) Co-management
Other: E-consult — In implementing the electronic consultation system in the private sector, the investigators will model the Expected Practice developed by the Los Angeles County Specialty-Primary Care Work Group. This eConsult system utilizes a "kickback" mechanism by which a specialist, who reviews the referral, can return it if it has not met certain baseline criteria (e.g. for a woman with OAB/urinary urgency: document negative UA, scheduled voids, titrate fluids to thirst, Kegels, antimuscarinics, optimize diuretic control, adjust any diuretics).
  Arms: Electronic Consult (E-consult)

SUMMARY:
The burden of urinary incontinence (UI) on American women is immense in both human and financial terms, and continues to rise with the aging US population. Although numerous non-surgical management strategies have proven efficacy for both stress and urge urinary incontinence, there remains a lack of appropriate UI management in the primary care setting. The goal of this multi-site cluster randomized comparative effectiveness trial is to compare the effects of two methods of nonsurgical UI care delivery - electronic consult vs. advanced practice provider (APP) co-management. These two evidence-based, practice-changing strategies are designed to improve the quality of care for an ethnically diverse population of women with UI, and, by reducing deficits in care, obtain better patient-reported outcomes. Both arms of the study will include basic physician education (academic detailing) and electronic clinical decision support. In Arm 1, the investigators will implement an electronic referral system (electronic referral), in which specialists will electronically review referrals and make additional recommendations if appropriate primary UI care was not provided. In Arm 2, Advanced Practice Provider (APP) co-management will reduce the burden of care on the PCPs by providing UI care, patient education, and assisting with patient self-management through dedicated televisits (APP co-management).

DETAILED DESCRIPTION:
The Burden of Urinary Incontinence on American Women is Immense: Although a great deal of research on quality of care has been conducted in many areas of medicine and surgery, there remains a relative paucity of data regarding the quality of care for women with urinary incontinence (UI). UI is defined by the International Continence Society as the complaint of any involuntary leakage of urine. The burden of UI on American women is immense in both human and financial terms, and continues to rise with the aging population. According to the National Health and Nutrition Examination Survey, the prevalence of UI among women ranges from 38%-53%. The lifetime risk of undergoing surgery for UI or pelvic organ prolapse is 20%. With the aging of the baby boomers it is projected that the number of women with UI will increase by 55% by 2050. UI negatively impacts health-related quality of life and is associated with embarrassment, stigma, and social isolation.

Primary Care Interventions for UI are Needed. In prior research by our team to provide background for the current proposal, the investigators sought to qualitatively assess challenges and barriers that primary care providers (PCPs) experience in caring for patients with UI. Twelve providers from the specialties of family medicine, general internal medicine, and geriatrics were interviewed. Providers described a lack of understanding of important components of a pelvic exam. Some male providers mentioned their own discomfort performing a pelvic exam on women. PCPs also discussed uncertainty in reaching a correct UI diagnosis (stress urinary incontinence, SUI, vs. urge urinary incontinence, UUI). There were also concerns about anticholinergic drug interactions and their association with cognitive impairment. There was a general lack of familiarity with medication options and dosing and a lack of knowledge about logistics in referring to pelvic floor physical therapy. Providers mentioned the need for an algorithm for the treatment of UI. They also described systems barriers included competing priorities with other medical issues, time limitations, and lack of interest in caring for patients with UI (unpublished).

The Care for Women with Urinary Incontinence Does Not Meet Recommended Standards of Care: With the assistance of co-I Dr. David Reuben, indicators of high quality were developed for vulnerable community-dwelling elders with urinary incontinence. Quality of care for UI was found to be grossly inadequate. In fact, pelvic examination, an important process measure, was performed in only 20% of older women with UI. Only 50% of patients received medical treatment for incontinence, and only 13% were prescribed behavioral modification, despite its proven effectiveness. In a sample of 247 women consecutively referred for new or worsening bothersome UI to FPMRS group practices at Cedars-Sinai, UCLA, and Harbor-UCLA, the investigators found that women ≥75 years of age were less likely than younger women to have received primary care for UI. In fact, older women were less likely to have a focused history obtained that differentiated between SUI and UUI (55% vs 77%, p<0.05), and were less likely to receive a pelvic exam (26% vs 50%, p<0.01) when compared to their younger counterparts. However, rates of behavioral management initiation were low in both older and younger groups, with only 30% of PCPs offering behavioral management (manuscript submitted to the American Journal of Medicine).

Access to Care for Underserved Latinas with Urinary Incontinence is Poor: Access to specialty care, which typically refers to in-person evaluation in a specialty clinic, is insufficient, particularly for underserved populations. Current physician shortages affect subspecialties disproportionately, and will be exacerbated as our population ages. In 2014, there were 3.6 million older adult Hispanics (8% of the older U.S. population); this number is expected to grow to 21.5 million by 2060 (data from the National Hispanic Council on Aging). Hispanic women bear a disproportionate burden of stress and mixed UI, yet may receive inferior care than other ethnic groups. The investigators conducted focus groups to compare perceptions and barriers between Spanish and English speaking women in public and private hospitals being treated for UI. Knowledge gaps were greater among Spanish speakers. Dr. Anger and her research team at UCLA-Olive View Medical Center (public hospital-based outpatient clinics) then sought to evaluate barriers in communication and disease understanding among office staff and interpreters when communicating with Spanish-speaking women with UI. Sixteen office staff and interpreters were interviewed. Patient-related barriers included a lack of understanding of anatomy and medical terminology and inhibited discussions due to embarrassment. Provider-related barriers included poor interpreter knowledge of pelvic floor vocabulary and the frequent use of office staff without interpreting credentials. This work identified obstacles in communication-barriers that only Spanish speaking women face. In this proposal the investigators seek to directly measure and improve the care provided to a heterogeneous population of women with UI, with the goals of improving care, improving UI outcomes, and improving knowledge and shared decision making, while simultaneously removing language barriers.

SIGNIFICANCE This study is significant for several reasons. First, in both study arms the investigators will bring subspecialty expertise to primary care settings, improving on interventions that have been done previously. The investigators will apply a set of QIs that represent the latest patient-centered outcomes research (PCOR) evidence regarding nonsurgical treatments for UI in women, and are all identifiable in the medical record. The QIs the investigators developed are a more comprehensive set than the original ACOVE indicators, developed by subspecialists and primary care providers. Whereas the ACOVE project focused on primary care interventions for UI among older adults at risk of decline, the new indicators distinguish stress vs. urge incontinence, are tailored for management of each type of incontinence, and are applicable across all populations of adult women. The research team's prior work has shown that, in a group of ambulatory patients aged 75+ who screened positive for UI (n=133), better quality of care for UI was associated with a measurable improvement in participant-reported outcomes. Composite quality scores (percentage of QIs passed per participant) and change in Incontinence Quality of Life (IQOL) questionnaire scores (range 0-100) were used as measurements. Each 10% increment in receipt of recommended care for UI was associated with a 1.4-point improvement in IQOL score (p=0.01), a clinically meaningful difference. The investigators expect to see a much larger impact on UI outcomes with this intervention, both arms of which have been tested and shown to make great strides in quality improvement.

There is abundant evidence supporting various nonsurgical management strategies for UI, including behavioral modification, pelvic floor exercises, and initiation of medication for overactive bladder/urge urinary incontinence. However, there are significant barriers to delivery of these strategies at the primary care level. The investigators have identified the two evidenced-based nonsurgical UI care delivery methods that have the greatest impact on care. One study arm to be evaluated is electronic co-management, which has multiple elements, all taken after the successful model created by the Los Angeles County Department of Health Services, the second largest public health care system in the country. eConsult (eConsult Health Ltd, London, England) is an electronic asynchronous consultation tool that was developed with the goals of increasing access, improving dialogue, optimizing efficiency, and enhancing primary care capacity. This infrastructure allows specialists to review electronic referrals and, when needed, return them and make recommendations to the PCP. This model empowers PCPs to more robustly manage conditions, and to streamline care if a specialist visit is necessary. The investigators will implement an electronic consultation system for patients in primary care offices at all sites. The investigators recently compared primary care for UI between private and public systems, and found that the public sector provided better primary care for UI.

The other study arm will be Advanced Practice Provider (APP) co-management. APPs will conduct the patient education portion of the intervention in the primary care setting. APP co-management has been shown to have a greater impact on quality than other educational measures for other chronic conditions affecting older persons, including dementia, and can substantially reduce the work needed on the part of PCPs. APP co-management will also leverage the recent Covid-19 related implementation of telemedicine. This will allow an APP to provide patient-centered care across different offices in a given healthcare system. In addition, based our prior findings of multiple levels of barriers to care for Spanish speaking women with UI, the research team will include certified bilingual APPs in the study so that Spanish speaking women will have a full understanding of what is taught to them. This will increase their knowledge level and allow for shared decision making (SDM) from a more informed perspective. Because UI is a chronic condition, patients need to play an active role in their care and be able to make their own decisions regarding UI management. Therefore, the investigators will also measure whether our intervention improves knowledge and perceived shared decision making. Lastly, the investigators will ensure that these approaches are tested in diverse populations to promote equitable care. As a secondary analysis, the investigators will test whether our proposed intervention reduces disparities in UI care. Should one, or even both, of our proposed interventions be effective in improving quality and outcomes, similar interventions can be easily implemented in most settings. Success of our intervention could lead to wide-scale implementation of effective, yet cost saving, quality improvement methods that reduce the burden of care on PCPs.

ELIGIBILITY:
Inclusion Criteria of Primary Care Physicians:

- Primary care physician belonging to a recruited office among one of three participating sites: UCSD, UCLA, KUMC

Inclusion Criteria of Patients:

* Age >18 y/o
* English or Spanish fluency
* Female
* Answers "yes" to incontinence screening tool and agrees to participate

Exclusion Criteria of Primary Care Physicians:

* Non-primary care specialty
* Does not belong to one of the participating offices

Exclusion Criteria of Patients:

* Age <18 y/o
* Answers "no" to incontinence screening tool and/or does not agree to participate
* Primary care provider (who reviews a list of patients that screen positive) deems patient ineligible due to pregnant, severe memory impairment, or psychiatric history preventing participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Provider Quality of Care - Evidence-Based Quality Indicators | Baseline
  Provider adherence to 13 evidence-based quality indicators will be compared across the E-Consult and Advanced Practice Provider (APP) Co-management arms.
Provider Quality of Care - Evidence-Based Quality Indicators | 6 months
  Provider adherence to 13 evidence-based quality indicators will be compared across the E-Consult and Advanced Practice Provider (APP) Co-management arms.
Change in provider quality of care measured by evidence-based quality indicators | Baseline, 6 months
  Provider adherence to 13 evidence-based quality indicators will be compared across the E-Consult and Advanced Practice Provider (APP) Co-management arms.

SECONDARY OUTCOMES:
Patient Symptoms - International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-SF) | Baseline
  The ICIQ-SF is a six item questionnaire that assesses the patient's frequency of urinary leakage and how it has negatively impacted their daily activities. The minimum ICIQ score of 0 indicates patient is not bothered by urinary incontinence, while the maximum ICIQ score of 21 indicates the patient's quality of life is negatively impacted a great deal by urinary incontinence.
Patient Symptoms - International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-SF) | 3 months
  The ICIQ-SF is a six item questionnaire that assesses the patient's frequency of urinary leakage and how it has negatively impacted their daily activities. The minimum ICIQ score of 0 indicates patient is not bothered by urinary incontinence, while the maximum ICIQ score of 21 indicates the patient's quality of life is negatively impacted a great deal by urinary incontinence.
Patient Symptoms - International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-SF) | 6 months
  The ICIQ-SF is a six item questionnaire that assesses the patient's frequency of urinary leakage and how it has negatively impacted their daily activities. The minimum ICIQ score of 0 indicates patient is not bothered by urinary incontinence, while the maximum ICIQ score of 21 indicates the patient's quality of life is negatively impacted a great deal by urinary incontinence.
Change in patients' urinary incontinence symptoms as measured by ICIQ-SF | Baseline, 3 months, 6 months
  The ICIQ-SF is a six item questionnaire that assesses the patient's frequency of urinary leakage and how it has negatively impacted their daily activities. The minimum ICIQ score of 0 indicates patient is not bothered by urinary incontinence, while the maximum ICIQ score of 21 indicates the patient's quality of life is negatively impacted a great deal by urinary incontinence.
Patient Symptoms - Urogenital Distress Inventory (UDI-6) | Baseline
  The UDI-6 is the urinary incontinence (UI) assessment tool endorsed by the American Urological Association and the Society for Urodynamics, Female Pelvic Medicine and Urogenital Reconstruction (SUFU). It contains only 6 questions and differentiates the type of UI (SUI vs. UUI), symptoms associated with UI, severity of symptoms and symptom bother. Furthermore, the UDI-6 gives a summative score that has been demonstrated to be sensitive to change with treatment and correlates with quality of life indices.
Patient Symptoms - Urinary symptoms as measured by Urogenital Distress Inventory (UDI-6) | 3 months
  The UDI-6 is the urinary incontinence (UI) assessment tool endorsed by the American Urological Association and the Society for Urodynamics, Female Pelvic Medicine and Urogenital Reconstruction (SUFU). It contains only 6 questions and differentiates the type of UI (SUI vs. UUI), symptoms associated with UI, severity of symptoms and symptom bother. Furthermore, the UDI-6 gives a summative score that has been demonstrated to be sensitive to change with treatment and correlates with quality of life indices.
Patient Symptoms - Urinary symptoms as measured by Urogenital Distress Inventory (UDI-6) | 6 months
  The UDI-6 is the urinary incontinence (UI) assessment tool endorsed by the American Urological Association and the Society for Urodynamics, Female Pelvic Medicine and Urogenital Reconstruction (SUFU). It contains only 6 questions and differentiates the type of UI (SUI vs. UUI), symptoms associated with UI, severity of symptoms and symptom bother. Furthermore, the UDI-6 gives a summative score that has been demonstrated to be sensitive to change with treatment and correlates with quality of life indices.
Change in patients' urinary symptoms as measured by UDI-6 | Baseline, 3 months, 6 months
  The UDI-6 is the urinary incontinence (UI) assessment tool endorsed by the American Urological Association and the Society for Urodynamics, Female Pelvic Medicine and Urogenital Reconstruction (SUFU). It contains only 6 questions and differentiates the type of UI (SUI vs. UUI), symptoms associated with UI, severity of symptoms and symptom bother. Furthermore, the UDI-6 gives a summative score that has been demonstrated to be sensitive to change with treatment and correlates with quality of life indices.
Patient Quality of Life - Incontinence Impact Questionnaire (IIQ-7) | Baseline
  The IIQ-7 is a seven-item questionnaire that assesses the impact of UI on health-related quality of life, with the minimum score of 0 indicating no impact and a maximum score of 21 indicating significant disruption of daily activities, relationships, and feelings.
Patient Quality of Life - Incontinence Impact Questionnaire (IIQ-7) | 3 months
  The IIQ-7 is a seven-item questionnaire that assesses the impact of UI on health-related quality of life, with the minimum score of 0 indicating no impact and a maximum score of 21 indicating significant disruption of daily activities, relationships, and feelings.
Patient Quality of Life - Incontinence Impact Questionnaire (IIQ-7) | 6 months
  The IIQ-7 is a seven-item questionnaire that assesses the impact of UI on health-related quality of life, with the minimum score of 0 indicating no impact and a maximum score of 21 indicating significant disruption of daily activities, relationships, and feelings.
Change in impact of UI on patients' quality of life as measure by the Incontinence Impact Questionnaire (IIQ-7) | Baseline, 3 months, 6 months
  The IIQ-7 is a seven-item questionnaire that assesses the impact of UI on health-related quality of life, with the minimum score of 0 indicating no impact and a maximum score of 21 indicating significant disruption of daily activities, relationships, and feelings.
Patient Decision Making - Shared Decision Making Questionnaire (SDM-Q-9) | 3 months
  Nine-item questionnaire that measures the extent to which patients are involved in the process of decision-making. This questionnaire requires patients to indicate how strongly they agree with given statements on a scale (completely disagree, strongly disagree, somewhat disagree, somewhat agree, strongly agree, completely agree).
Patient Satisfaction - Net Promoter Score | 3 months
  The Net Promoter Score evaluates a patient's willingness to refer a friend to the provider from whom they received care and to the institution where they received care. Patients respond on a 5-item Likert score on how likely they would be to make the referrals. Patients are ranked as "Detractors", "Passive", and "Promoters". The Net Promoter Score is calculated by subtracting the group percentage of "Promoters" from the group percentage of "Detractors."
Patient Knowledge - Pelvic Floor Awareness and Knowledge Survey (P-FAKS) | Baseline
  Thirty-one-item questionnaire assessing patient knowledge in three domains: POP (11 items), SUI (10 items) and OAB (10 items) with questions on condition pathophysiology, management, and quality of life.
Patient Knowledge - Pelvic Floor Awareness and Knowledge Survey (P-FAKS) | 6 months
  Thirty-one-item questionnaire assessing patient knowledge in three domains: POP (11 items), SUI (10 items) and OAB (10 items) with questions on condition pathophysiology, management, and quality of life.
Change in patients' knowledge as measured by the P-FAKS | Baseline, 6 months
  Thirty-one-item questionnaire assessing patient knowledge in three domains: POP (11 items), SUI (10 items) and OAB (10 items) with questions on condition pathophysiology, management, and quality of life.
Provider Knowledge - Pelvic Floor Awareness and Knowledge Survey (P-FAKS) | Baseline
  Nine-item questionnaire that measures the extent to which patients are involved in the process of decision-making. This questionnaire requires patients to indicate how strongly they agree with given statements on a scale (completely disagree, strongly disagree, somewhat disagree, somewhat agree, strongly agree, completely agree).
Provider Knowledge - Pelvic Floor Awareness and Knowledge Survey (P-FAKS) | 6 months
  Thirty-one-item questionnaire assessing patient knowledge in three domains: POP (11 items), SUI (10 items) and OAB (10 items) with questions on condition pathophysiology, management, and quality of life.
Change in provider knowledge as measured by the P-FAKS | Baseline, 6 months
  Thirty-one-item questionnaire assessing patient knowledge in three domains: POP (11 items), SUI (10 items) and OAB (10 items) with questions on condition pathophysiology, management, and quality of life.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California Los Angeles, Los Angeles, California
  - University of California San Diego, San Diego, California
  - University of Kansas, Lawrence, Kansas

IPD SHARING:
Plan to Share IPD: Yes
Available by request.

REFERENCES:
- [Background] Dieter AA, Wilkins MF, Wu JM. Epidemiological trends and future care needs for pelvic floor disorders. Curr Opin Obstet Gynecol. 2015 Oct;27(5):380-4. doi: 10.1097/GCO.0000000000000200. PMID 26308198
- [Background] Anger JT, Scott VC, Kiyosaki K, Khan AA, Weinberg A, Connor SE, Roth CP, Wenger N, Shekelle P, Litwin MS. Development of quality indicators for women with urinary incontinence. Neurourol Urodyn. 2013 Nov;32(8):1058-63. doi: 10.1002/nau.22353. Epub 2013 Sep 16. PMID 24105879
- [Background] Anger JT, Alas A, Litwin MS, Chu SD, Bresee C, Roth CP, Rashid R, Shekelle P, Wenger NS. The Quality of Care Provided to Women with Urinary Incontinence in 2 Clinical Settings. J Urol. 2016 Oct;196(4):1196-200. doi: 10.1016/j.juro.2016.05.005. Epub 2016 May 7. PMID 27164512
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Background] Anger JT, Saigal CS, Litwin MS; Urologic Diseases of America Project. The prevalence of urinary incontinence among community dwelling adult women: results from the National Health and Nutrition Examination Survey. J Urol. 2006 Feb;175(2):601-4. doi: 10.1016/S0022-5347(05)00242-9. PMID 16407004
- [Background] Markland AD, Richter HE, Fwu CW, Eggers P, Kusek JW. Prevalence and trends of urinary incontinence in adults in the United States, 2001 to 2008. J Urol. 2011 Aug;186(2):589-93. doi: 10.1016/j.juro.2011.03.114. PMID 21684555
- [Background] Wu JM, Hundley AF, Fulton RG, Myers ER. Forecasting the prevalence of pelvic floor disorders in U.S. Women: 2010 to 2050. Obstet Gynecol. 2009 Dec;114(6):1278-1283. doi: 10.1097/AOG.0b013e3181c2ce96. PMID 19935030
- [Background] Mesens T, Aich A, Bhal PS. Late erosions of mid-urethral tapes for stress urinary incontinence--need for long-term follow-up? Int Urogynecol J Pelvic Floor Dysfunct. 2007 Sep;18(9):1113-4. doi: 10.1007/s00192-007-0301-4. Epub 2007 Mar 9. PMID 17347793
- [Background] Schnelle JF, Smith RL. Quality indicators for the management of urinary incontinence in vulnerable community-dwelling elders. Ann Intern Med. 2001 Oct 16;135(8 Pt 2):752-8. doi: 10.7326/0003-4819-135-8_part_2-200110161-00015. No abstract available. PMID 11601959
- [Background] Gnanadesigan N, Saliba D, Roth CP, Solomon DH, Chang JT, Schnelle J, Smith R, Shekelle PG, Wenger NS. The quality of care provided to vulnerable older community-based patients with urinary incontinence. J Am Med Dir Assoc. 2004 May-Jun;5(3):141-6. doi: 10.1097/01.JAM.0000123026.47700.1A. PMID 15115573
- [Background] Bisgaier J, Rhodes KV. Auditing access to specialty care for children with public insurance. N Engl J Med. 2011 Jun 16;364(24):2324-33. doi: 10.1056/NEJMsa1013285. PMID 21675891
- [Background] Rhodes KV, Bisgaier J, Lawson CC, Soglin D, Krug S, Van Haitsma M. "Patients who can't get an appointment go to the ER": access to specialty care for publicly insured children. Ann Emerg Med. 2013 Apr;61(4):394-403. doi: 10.1016/j.annemergmed.2012.10.030. Epub 2013 Jan 8. PMID 23312670
- [Background] Mehrotra A, Forrest CB, Lin CY. Dropping the baton: specialty referrals in the United States. Milbank Q. 2011 Mar;89(1):39-68. doi: 10.1111/j.1468-0009.2011.00619.x. PMID 21418312
- [Background] Dall TM, Gallo PD, Chakrabarti R, West T, Semilla AP, Storm MV. An aging population and growing disease burden will require a large and specialized health care workforce by 2025. Health Aff (Millwood). 2013 Nov;32(11):2013-20. doi: 10.1377/hlthaff.2013.0714. PMID 24191094
- [Background] McKibben MJ, Kirby EW, Langston J, Raynor MC, Nielsen ME, Smith AB, Wallen EM, Woods ME, Pruthi RS. Projecting the Urology Workforce Over the Next 20 Years. Urology. 2016 Dec;98:21-26. doi: 10.1016/j.urology.2016.07.028. Epub 2016 Aug 1. PMID 27491965
- [Background] Alas AN, Dunivan GC, Wieslander CK, Sevilla C, Barrera B, Rashid R, Maliski S, Eilber K, Rogers RG, Anger JT. Health Care Disparities Among English-Speaking and Spanish-Speaking Women With Pelvic Organ Prolapse at Public and Private Hospitals: What Are the Barriers? Female Pelvic Med Reconstr Surg. 2016 Nov/Dec;22(6):460-466. doi: 10.1097/SPV.0000000000000315. PMID 27636216
- [Background] Khan AA, Sevilla C, Wieslander CK, Moran MB, Rashid R, Mittal B, Maliski SL, Rogers RG, Anger JT. Communication barriers among Spanish-speaking women with pelvic floor disorders: lost in translation? Female Pelvic Med Reconstr Surg. 2013 May-Jun;19(3):157-64. doi: 10.1097/SPV.0b013e318288ac1c. PMID 23611934
- [Background] Min LC, Reuben DB, Adams J, Shekelle PG, Ganz DA, Roth CP, Wenger NS. Does better quality of care for falls and urinary incontinence result in better participant-reported outcomes? J Am Geriatr Soc. 2011 Aug;59(8):1435-43. doi: 10.1111/j.1532-5415.2011.03517.x. Epub 2011 Aug 1. PMID 21806560
- [Background] Barnett ML, Yee HF Jr, Mehrotra A, Giboney P. Los Angeles Safety-Net Program eConsult System Was Rapidly Adopted And Decreased Wait Times To See Specialists. Health Aff (Millwood). 2017 Mar 1;36(3):492-499. doi: 10.1377/hlthaff.2016.1283. PMID 28264951
- [Background] Soni SM, Giboney P, Yee HF Jr. Development and Implementation of Expected Practices to Reduce Inappropriate Variations in Clinical Practice. JAMA. 2016 May 24-31;315(20):2163-4. doi: 10.1001/jama.2016.4255. No abstract available. PMID 27218624
- [Background] Jennings LA, Tan Z, Wenger NS, Cook EA, Han W, McCreath HE, Serrano KS, Roth CP, Reuben DB. Quality of Care Provided by a Comprehensive Dementia Care Comanagement Program. J Am Geriatr Soc. 2016 Aug;64(8):1724-30. doi: 10.1111/jgs.14251. Epub 2016 Jun 29. PMID 27355394
- [Background] Bordeianou LG, Anger JT, Boutros M, Birnbaum E, Carmichael JC, Connell KA, De EJB, Mellgren A, Staller K, Vogler SA, Weinstein MM, Yafi FA, Hull TL; Members of the Pelvic Floor Disorders Consortium Working Groups on Patient-Reported Outcomes. Measuring Pelvic Floor Disorder Symptoms Using Patient-Reported Instruments: Proceedings of the Consensus Meeting of the Pelvic Floor Consortium of the American Society of Colon and Rectal Surgeons, the International Continence Society, the American Urogynecologic Society, and the Society of Urodynamics, Female Pelvic Medicine and Urogenital Reconstruction. Female Pelvic Med Reconstr Surg. 2020 Jan/Feb;26(1):1-15. doi: 10.1097/SPV.0000000000000817. No abstract available. PMID 31833996
- [Background] McGlynn EA, Asch SM, Adams J, Keesey J, Hicks J, DeCristofaro A, Kerr EA. The quality of health care delivered to adults in the United States. N Engl J Med. 2003 Jun 26;348(26):2635-45. doi: 10.1056/NEJMsa022615. PMID 12826639
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Min LC, Reuben DB, MacLean CH, Shekelle PG, Solomon DH, Higashi T, Chang JT, Roth CP, Kamberg CJ, Adams J, Young RT, Wenger NS. Predictors of overall quality of care provided to vulnerable older people. J Am Geriatr Soc. 2005 Oct;53(10):1705-11. doi: 10.1111/j.1532-5415.2005.53520.x. PMID 16181169